CLINICAL TRIAL: NCT00773253
Title: Pre-injection, Multi-channel EMG Mapping to Optimize Botulinum Toxin Type A Efficacy in Cervical Dystonia.
Brief Title: Botox for Cervical Dystonia Following EMG Mapping
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Allergan cervical dystonia
Record Dates: First submitted 2008-10-14; First posted 2008-10-16 (Estimated); Results first posted 2011-10-13 (Estimated); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Cervical Dystonia
Keywords: dystonia; cervical dystonia; Botox; idiopathic primary cervical dystonia
MeSH Terms: conditions — Torticollis; Dystonia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard EMG-guided Botox injection (Active Comparator): All patients will undergo injection using conventional single channel EMG-guided technique. This will be used as a baseline for multi-channel mapping-based injections. Patients will be randomized to undergo single-channel vs. multi-channel assessment upon study entry and will then cross over to the alternate arm.
  Interventions: Drug: Botulinum toxin A
- Multi-channel EMG-guided Botox injection (Experimental): Patients will receive multi-channel EMG-guided Botox injection before or after they have been treated with single-channel EMG-guided Botox, depending on which group they are assigned in the cross-over design.
  Interventions: Drug: Botulinum toxin A

INTERVENTIONS:
Drug: Botulinum toxin A — All patients will be treated with Botox using both single-channel and multi-channel EMG mapping.
  Other Names: Botox

SUMMARY:
The purpose of this study is to determine how to improve treatment of patients with cervical dystonia who have not been helped with standard Botox injections. This study is for patients with cervical dystonia who have not benefited from treatment with Botox using conventional "single lead electromyographic (EMG) techniques" for injection. The study aim is to see if these patients may have significantly more benefit if their Botox is injected into muscles that have been chosen with a multi-channel EMG mapping study of the neck prior to Botox injection.

DETAILED DESCRIPTION:
The most common type of primary late-onset dystonia is cervical dystonia. Botulinum toxin A (BTX-A) injections are a safe and effective treatment for cervical dystonia in a majority of patients, however, a significant minority of patients (between 15 and 25%) have a suboptimal response to Botulinum toxin therapy. It is unclear why some patients do not respond maximally to neurotoxin therapy.

Studies using needle electromyographic "mapping" in the evaluation of cervical dystonia have revealed that clinical examination alone is insufficient for determining which muscles contribute to the dystonic movement. When compared to needle electromyography (EMG) "mapping studies", experienced movement disorders specialists correctly identify only 59% of active muscles and believe that 25% of muscles which upon EMG evaluation are found to be quiescent, are involved in the dystonia. The selection of incorrect muscles for injection of Botulinum toxin may explain why some patients have a sub-optimal response.

This study seeks to measure outcomes when the muscles involved in dystonia are identified using "mapping" via an 8-12 channel EMG. In the proposed study, the most involved/active dystonic muscles will be correctly identified through simultaneous 8-12 channel mapping resulting in a more informed injection strategy, which may improve response to Botulinum toxin A treatment as compared to single lead EMG based injections. This study changes routine clinical care only by adding the step of studying the muscles of the neck with simultaneous EMG mapping to allow a more objective injection strategy.

ELIGIBILITY:
Inclusion criteria:

* Male or female subjects, 18 to 75 years of age.
* Ability to follow study instructions and complete all required visits.
* Subject meets diagnostic criteria for idiopathic primary cervical dystonia.
* Subject has at least moderate severity Cervical Dystonia, with a baseline rating of at least 30 on the total TWSTRS and at least 15 on the TWSTRS motor severity subsection.
* Patients have had a suboptimal response to 2 previous Botulinum toxin injections at an outside facility.
* Patients will not have received Botulinum toxin within 16 weeks of the start of the study.
* In order to not confound the clinical response to BTX-A injections, all patients enrolled must have been on a stable medication regimen for 30 days. If they are not on medication at the initiation of the study, they will not be started on medication. Patients must be on the same medication regimen through the entire study including assessment of both single lead EMG based injections and "mapping" based injections. Medications cannot be stopped during the study to avoid confounding the clinical response to BTX-A.

Exclusion Criteria:

* Known allergy or sensitivity to any of the components in BTX-A.
* Uncontrolled clinically significant medical condition other than the condition under evaluation
* Females with a positive pregnancy test, or who are breast-feeding, planning a pregnancy during the study, who think that they may be pregnant at the start of the study or females of childbearing potential who are unable or unwilling to use a reliable form of contraception during the study.
* Participation in another medication or device study or within 3 months of enrollment in this study.
* Patients know to have a positive frontalis test or have previously tested positive for the presence of BTX-A antibodies will be excluded.
* Any known evidence of cervical contractures or significant spinal deformity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-04; Primary Completion 2010-10 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graham A. Glass, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard EMG Guided Injections Then Multi-channel Injections: All patients will undergo injection using conventional single channel (standard)EMG-guided technique. This will be used as a baseline for multi-channel mapping-based injections. Patients will be randomized to undergo single-channel vs. multi-channel assessment upon study entry and will then cross over to the alternate arm.
- Multi-channel EMG-guided Botox Injection Then Standard EMG Inj: Patients will receive multi-channel EMG-guided Botox injection before or after they have been treated with single-channel (standard) EMG-guided Botox, depending on which group they are assigned in the cross-over design.
Period: First Intervention (Week 0-24)
Arm/Group | Standard EMG Guided Injections Then Multi-channel Injections | Multi-channel EMG-guided Botox Injection Then Standard EMG Inj
Started | 5 | 5
Completed | 5 | 4
Not Completed | 0 | 1
Not completed — Frontalis Test Negative | 0 | 1
Period: Second Intervention (Week 24-48)
Arm/Group | Standard EMG Guided Injections Then Multi-channel Injections | Multi-channel EMG-guided Botox Injection Then Standard EMG Inj
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard EMG Guided Injections Then Multi-channel: All patients will undergo injection using conventional single channel EMG-guided technique. This will be used as a baseline for multi-channel mapping-based injections. Patients will be randomized to undergo single-channel vs. multi-channel assessment upon study entry and will then cross over to the alternate arm.
- Multi-channel EMG-guided Botox Injection Then Single Channel: Patients will receive multi-channel EMG-guided Botox injection before or after they have been treated with single-channel EMG-guided Botox, depending on which group they are assigned in the cross-over design.
- Total: Total of all reporting groups
Arm/Group | Standard EMG Guided Injections Then Multi-channel | Multi-channel EMG-guided Botox Injection Then Single Channel | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (5.2) | 54.7 (5.1) | 55.4 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Pre- and Post-injection Toronto Western Spasmodic Torticollis Rating Scale(TWSTRS): Global Clinical Impression Scale (GCI); Visual Analog Scale(VAS)
Time Frame: pre-injection, week 16, 20, 36, and 40
Population: PI left institution. Efforts to contact PI to obtain data have been unsuccessful.
Arm/Group | Standard EMG-guided Botox Injection | Multi-channel EMG-guided Botox Injection
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Mean Percentage Change in Total Toronto Western Spasmodic Torticollis Rating Scale
Description: Mean Percentage change in Toronto Western Spasmodic Torticollis Rating Scale. This scale ranges from 0 (normal) to 85 (very severe).
Time Frame: baseline and 48 weeks
Population: All participants that completed all phases of the study
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Standard EMG Guided Injections: All patients underwent single channel (standard)EMG-guided technique.
- Multi-channel EMG-guided Botox Injection: Patients will receive multi-channel EMG-guided Botox injection.
Arm/Group | Standard EMG Guided Injections | Multi-channel EMG-guided Botox Injection
Number analyzed (Participants) | 9 | 9
percent change | 9 (20.8) | 23.5 (15.7)

ADVERSE EVENTS:
Arm/Group | Standard EMG Guided Injections | Multi-channel EMG-guided Botox Injection
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10

LIMITATIONS AND CAVEATS:
One patient received single channel injection, but did not get multi-channel injection because the frontalis test showed immunity to botulinum toxin indicating no possibility of clinical benefit. This is an exclusion criterion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No